CLINICAL TRIAL: NCT02187341
Title: Effects of Exercise and 5-HTP on Cortisol Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benedictine University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Ben-0614b
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Plasma Cortisol
MeSH Terms: interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-HTP (Experimental): 200 mg 5-HTP capsule will be ingested 2h prior to reporting to the laboratory.
  Interventions: Dietary Supplement: 5-HTP
- Placebo (Placebo Comparator): For these visit subjects will ingest placebo (Sugar pill) capsule 2 hours before reporting to the laboratory.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 5-HTP — Volunteers participate in two visits at least 5 days apart . The day of their visit they ingest (2 hours before reporting to the laboratory) either a capsule containing 200 mg of 5-HTP or a capsule containing placebo (sugar pill). The order of the visits is randomized
  Arms: 5-HTP
Dietary Supplement: Placebo — Volunteers participate in two visits at least 5 days apart . The day of their visit they ingest (2 hours before reporting to the laboratory) either a capsule containing 200 mg of 5-HTP or a capsule containing placebo (sugar pill). The order of the visits is randomized
  Arms: Placebo

SUMMARY:
It has been shown that 5-HTP stimulates cortisol levels in plasma and saliva. Similarly, it has been shown that intense exercise stimulates an increase in plasma and salivary cortisol levels. The purpose of this study is to examine the combined effects of 5-HTP + intense exercise on plasma and salivary cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, not taking medication known to alter glucocorticoid metabolism

Exclusion Criteria:

* Diabetes
* Obesity
* Hypertension
* Coronary artery disease
* Psychiatric disorders
* Any disease preventing them from participating in intense exercise
* Subjects taking medication known to interfere with glucocorticoid metabolism will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma cortisol from baseline to 20 minutes post | baseline, 20 min
  Plasma cortisol will be assessed at baseline and 20 min post exercise and compared to baseline, and compared between treatments: 5-HTP vs placebo visit. The interventions are acute ( 1 dose, 1 day), for 5-HTP and for placebo, there is no follow up. The interventions are at least 1 week apart. For a given subject, the estimated time for study completion for the 2 treatments is 10 to 30 days

SECONDARY OUTCOMES:
Change in plasma cortisol from baseline to 5 minutes post | baseline, 5 minutes
  Plasma cortisol will be assessed at baseline and 5 min post exercise and compared to baseline, and compared between treatments: 5-HTP vs placebo visit. The interventions are acute ( 1 dose, 1 day), for 5-HTP and for placebo, there is no follow up. The interventions are at least 1 week apart. For a given subject, the estimated time for study completion for the 2 treatments is 10 to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Del Corral, PhD-MD, Principal Investigator — Benedictine University
Locations (1):
- Benedictine University, Lisle, Illinois, United States